CLINICAL TRIAL: NCT07157683
Title: Biomarkers in Systemic Histiocytosis
Acronym: Bio-Histio
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250660
Record Dates: First submitted 2025-07-23; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: Systemic Histiocytosis (Disorder)
Keywords: histiocytosis
MeSH Terms: conditions — Histiocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — - If a blood sample is drawn as part of standard care, up to six additional EDTA tubes (42 mL max) will be collected for research.
  In addition, the following optional samples may be collected, depending on investigator assessment and/or patient preference:
  * Saliva sample (if no blood draw is performed)
  * Urine sample
  * Stool sample"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biospecimen collection — If a blood sample is drawn as part of standard care, up to six additional EDTA tubes (42 mL max) will be collected for research.
  In addition, the following optional samples may be collected, depending on investigator assessment and/or patient preference:
  * Saliva sample (if no blood draw is performed)
  * Urine sample
  * Stool sample"

SUMMARY:
Systemic histiocytoses in adults (Langerhans cell histiocytosis, Erdheim-Chester disease, and Rosai-Dorfman disease) are rare inflammatory disorders in which recent discoveries have identified a clonal origin, with activating mutations in the MAP kinase pathway, enabling access to targeted therapies. However, the mechanism by which these mutations induce an inflammatory profile in tissue histiocytes remains largely unknown.

Despite these advances, there is a clear need to refine diagnostic and prognostic classification, to identify the biological mechanisms involved in the onset and progression of these diseases, to develop new targeted strategies, and to establish minimally invasive monitoring methods (liquid biopsies).

This project aims to make a decisive contribution toward these goals.

DETAILED DESCRIPTION:
Systemic histiocytoses are rare diseases with a clinical spectrum ranging from mild forms to severe, life-threatening multi-organ involvement. Numerous recent studies have identified somatic mutations in the MAP kinase pathway in tissue-infiltrating histiocytes, providing a better understanding of the disease pathophysiology and enabling access to more effective targeted therapies. However, due to the extreme rarity of these diseases, many unknowns remain.

These mutations do not appear to induce a proliferative oncogenic process, as seen in cancers where similar mutations have been identified. Instead, they seem to trigger a pro-inflammatory and pro-fibrotic immune response, ultimately leading to organ damage. The immune mechanisms induced by these mutations in histiocytes remain unexplored.

There are also currently no reliable data to accurately predict disease progression, including survival, treatment response, remission, or organ involvement.

It is therefore essential to establish patient cohorts to improve disease understanding and to identify effective diagnostic, prognostic, and predictive biomarkers-whether for standard treatment response or as potential theranostic markers (actionable by a specific treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient followed for systemic histiocytosis in Internal Medicine Department 2 at Pitié-Salpêtrière Hospital
* Non-opposition to participation in the study

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients without French social security or covered by State Medical Aid (AME)
* Patients deprived of liberty by judicial or administrative decision, or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with systemic histiocytosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2040-10-01 (Estimated); Study Completion 2040-10-01 (Estimated)

PRIMARY OUTCOMES:
Identification of new biomarkers involved in histiocytosis | 10 years
  Plasma concentrations of several cytokines and chemokines involved in inflammation and fibrosis will be assessed using ELISA and Luminex assays (CSF, EGF, GM-CSF, FGF-basic, IFN-α, MCP-1, HGF, IFN-γ, MIG, VEGF, IL-1β, MIP-1α, IL-1RA, MIP-1β, IL-2, RANTES, IL-2R, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p40/p70), IL-13, IL-15, IL-17, TNF-α, and Eotaxin),

SECONDARY OUTCOMES:
Identification of new biomarkers involved in histiocytosis | 10 years
  using targeted transcriptomic profiling: total RNAseq using the Human Immunology v2 panel (Nanostring, 594 genes),
Identification of new biomarkers involved in histiocytosis | 10 years
  using single-cell RNA sequencing
Identification of new biomarkers involved in histiocytosis | 10 years
  using flow cytometry and mass cytometry analyses of 37 immune cell subsets using a dedicated 30-marker panel.
Description of the correlation between the identified biomarkers and clinical manifestation of histiocytosis | 10 years
Description of the correlation between the identified biomarkers and prognosis of histiocytosis | 10 years
  like mortality, or organ damage
Description of the correlation between the identified biomarkers and response to treatment | 10 years
  complete response, partial response, stable disease, disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Department 2 at Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.